CLINICAL TRIAL: NCT00673660
Title: Assessment Of Statin Treatment Compliance In Dyslipidemia Patients: An Observational Study
Brief Title: Observational Study On Compliance Of Statin Treatment Of Patients With High Blood Cholesterol Levels
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A2581156
Record Dates: First submitted 2008-05-01; First posted 2008-05-07 (Estimated); Results first posted 2010-11-04 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Dyslipidemia
Keywords: Statins; Compliance; Dyslipidemia
MeSH Terms: conditions — Dyslipidemias; Patient Compliance | interventions — Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimen is retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Statins: Patients with dyslipidemia who are taking or planning to take a statin treatment (Atorvastatin, Fluvastatin, Prevastatin, Rosuvastatin, Simvastatin or generics).
  Interventions: Behavioral: Patient Compliance

INTERVENTIONS:
Behavioral: Patient Compliance — Compliance of patients to statin treatment and reasons of compliance or non compliance will be obtained by Patient Reported Outcomes (PROs) every 3 months.

SUMMARY:
The purpose of the study is to show the compliance rates of the patients to statin treatment and the reasons of non-compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with dyslipidemia and taking or planning to take statin treatment.
* Patients living in the same city of the study center. o Patients aged 18 years and over.

Exclusion Criteria:

* Patients with severe systemic disease
* Patients with alcohol and drug addiction and/or mental disease
* Patients nursing or pregnant, or planning to get pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with dyslipidemia and taking or planning to take statin treatment. Patients living in the same city of the study center. Patients aged 18 years old and over.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Turkey (Türkiye) (4):
  - Pfizer Investigational Site, Mecidiyeköy, Istanbul
  - Pfizer Investigational Site, Bolu
  - Pfizer Investigational Site, Haseki/Istanbul
  - Pfizer Investigational Site, Istanbul

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581156&StudyName=Observational%20Study%20On%20Compliance%20Of%20Statin%20Treatment%20Of%20Patients%20With%20High%20Blood%20Cholesterol%20Levels

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational study evaluating compliance to statin treatment in participants with dyslipidemia. Data available at each visit was recorded in case report forms (CRFs). No laboratory measurements were performed. The gender of 2 subjects was not recorded.
Groups:
- Statins: Participants with dyslipidemia who were taking or were planning to take a statin treatment (Atorvastatin, Fluvastatin, Prevastatin, Rosuvastatin, Simvastatin, or generics).
Period: Overall Study
Arm/Group | Statins
Started | 375
Completed | 268
Not Completed | 107
Not completed — Lost to Follow-up | 107

BASELINE CHARACTERISTICS:
Arm/Group | Statins
Number analyzed (Participants) | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (10.6)
Sex/Gender, Customized [Number; unit: participants]
  Female | 186
  Male | 187
  Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Compliant With Statin Treatment
Description: The physician asked participants about their compliance with medication use, which was defined as not skipping or forgetting dosing or not delaying the dosing time at least 80 percent (%) of the days in which the medication was used.
Time Frame: Month 12
Population: Primary analysis population: participants diagnosed with dyslipidemia who were taking or planning to take statin treatment. Subset of evaluable participants were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Statins
Number analyzed (Participants) | 375
Percentage of participants | 86.7

2. Secondary Outcome: Available Lipid Profiles of Compliant and Non-compliant Participants
Description: Available laboratory measurements of participants were recorded in CRFs.
Time Frame: Month 12
Population: Primary analysis population, subset of evaluable participants.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Groups:
- Compliant With Statin Treatment: Participants with dyslipidemia who were compliant with statin treatment (Atorvastatin, Fluvastatin, Prevastatin, Rosuvastatin, Simvastatin, or generics).
- Non-compliant With Statin Treatment: Participants with dyslipidemia who were non-compliant with statin treatment (Atorvastatin, Fluvastatin, Prevastatin, Rosuvastatin, Simvastatin, or generics).
Arm/Group | Compliant With Statin Treatment | Non-compliant With Statin Treatment
Number analyzed (Participants) | 228 | 35
milligrams per deciliter
  Total cholesterol | 178.94 (41.17) | 231.59 (45.89)
  Low Density Lipoprotein (LDL) cholesterol | 101.61 (33.50) | 156.48 (41.22)
  High Density Lipoprotein (HDL) cholesterol | 50.70 (14.47) | 53.33 (23.76)
  Triglyceride | 137.80 (70.24) | 156.89 (65.32)
Statistical Analysis 1: Comparison: Compliant With Statin Treatment vs Non-compliant With Statin Treatment; Total cholesterol; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-Values less than 0.05 were considered statistically significant
Statistical Analysis 2: Comparison: Compliant With Statin Treatment vs Non-compliant With Statin Treatment; LDL cholesterol; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-Values less than 0.05 were considered statistically significant
Statistical Analysis 3: Comparison: Compliant With Statin Treatment vs Non-compliant With Statin Treatment; HDL cholesterol; Test type: Superiority or Other; p = 0.972, t-test, 1 sided — p-Values less than 0.05 were considered statistically significant
Statistical Analysis 4: Comparison: Compliant With Statin Treatment vs Non-compliant With Statin Treatment; Triglycerides; Test type: Superiority or Other; p = 0.034, t-test, 2 sided — p-Values less than 0.05 were considered statistically significant

3. Secondary Outcome: Number of Participants With Reasons of Compliance to Statin Treatment
Description: Compliance with medication use defined as not skipping or forgeting dosing or not delaying the dosing time at least 80 percent (%) of the days in which the medication was used. Participants were called for a final visit . Compliance with drug dosage was recorded.
Time Frame: Month 12
Population: Primary analysis population. The number of participants with reasons of compliance to statin treatment were not collected or analyzed.
Arm/Group | Statins
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Reasons of Non-compliance to Statin Treatment
Description: Participants were called for a final visit and reasons for non-compliance were recorded.
Time Frame: Month 12
Population: Primary analysis population, subset of evaluable participants
Measure: Number; unit: participants
Arm/Group | Statins
Number analyzed (Participants) | 268
participants
  Lab parameters were normal in final assessment | 11
  Difficulty obtaining prescribed drugs | 8
  Forgot to take drug | 7
  Don't like taking drugs | 9
  Thought it not necessary to take drug | 5
  Was late in taking drug | 1
  Don't think it necesary to take drug continuously | 0
  Don't want to use drugs for a long time | 4
  Experienced adverse events (AEs) | 3
  Think they are useless | 0
  Afraid of becoming an addict | 2
  I am resting my liver | 0
  Can't take drugs regularly due to high drug price | 1
  Other | 9

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Statins at Visit 2; Statins at Visit 3; Statins at Visit 4; Statins Visit 5: Participants with dyslipidemia who were taking or were planning to take a statin treatment (Atorvastatin, Fluvastatin, Prevastatin, Rosuvastatin, Simvastatin, or generics).
Arm/Group | Statins at Visit 2 | Statins at Visit 3 | Statins at Visit 4 | Statins Visit 5
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/76 | 0/44 | 0/268
Other Adverse Events (participants affected / at risk) | 5/153 | 4/76 | 4/44 | 6/268
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Statins at Visit 2 (N=153) | Statins at Visit 3 (N=76) | Statins at Visit 4 (N=44) | Statins Visit 5 (N=268)
Headache (General disorders) | 1 | 0 | 0 | 1
Back pain (General disorders) | 1 | 1 | 1 | 0
Allergic reaction (General disorders) | 1 | 1 | 0 | 0
Arthralgia (General disorders) | 1 | 1 | 0 | 0
Myalgia (General disorders) | 0 | 0 | 0 | 1
Dizziness (General disorders) | 1 | 0 | 0 | 1
Constipation (General disorders) | 0 | 0 | 0 | 1
Dyspepsia (General disorders) | 0 | 0 | 1 | 0
Nausea (General disorders) | 2 | 0 | 0 | 0
Gas (General disorders) | 2 | 0 | 0 | 0
Pharyngitis (General disorders) | 0 | 0 | 1 | 0
Elevated liver enzyme levels (General disorders) | 1 | 2 | 1 | 1
Rash on hands (General disorders) | 0 | 1 | 0 | 0
Cough (General disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (General disorders) | 0 | 0 | 1 | 0
Visual impairment (General disorders) | 0 | 0 | 0 | 1
Renal failure (General disorders) | 0 | 0 | 0 | 1
Vertigo (General disorders) | 0 | 0 | 0 | 1
Other (General disorders) | 3 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The registered endpoint - observing reasons of compliance or non-compliance to statin treatment - was separated into outcome measure 6 and 7 because observing reasons for compliance with statin treatment were not collected or analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.